CLINICAL TRIAL: NCT06573632
Title: Does Perioperative Parenteral Nutrition Affect Outcome in Patients Undergoing Major Abdominal Surgeries
Brief Title: Perioperative TPN Improves Surgical Outcomes
Status: Completed | Type: Observational
Sponsor: Nepal Medical College and Teaching Hospital (Other)
Responsible Party: Principal Investigator, Nabin Pokharel, Prof Dr. Nabin Pokharel, Head of Department of Surgical Gastroenterology, Nepal Medical College and Teaching Hospital
Other Study IDs: 26-079/080
Record Dates: First submitted 2024-08-15; First posted 2024-08-27 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Parenteral Nutrition; Major Surgery; Malnutrition
Keywords: parenteral nutrition; TPN; major surgery; malnutrition in surgery; clavien-dindo classification
MeSH Terms: conditions — Hyperphagia; Malnutrition

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Malnutrition: All malnutrition patients to received TPN for 5 days preoperatively as applicable and continued postoperatively.
  Interventions: Dietary Supplement: TPN-N7 Baxter

INTERVENTIONS:
Dietary Supplement: TPN-N7 Baxter — providing TPN to all malnutrition patients preoperatively as well as postoperatively.

SUMMARY:
Preoperative optimization of patients is a well known concept. Not all patients can tolerate feeds and as such TPN is given. TPN given preoperatively and continued postoperatively in selected group of patients can significantly improve the surgical outcomes and lower the morbidity as well as mortality. So the investigators aim to find the impact of TPN in malnutritional surgical patients.

DETAILED DESCRIPTION:
Any patient who is at risk of malnutrition as well as already malnutritioned were given preoperative TPN for 5 days. After 5 days, elective surgery was done and TPN was continued postoperatively until patient could consume 50% of their daily requirements orally. Patients who underwent emergency surgeries were also enrolled in this study as these patients could receive TPN only postoperatively.

Daily patient charting with Clavien Dindo Classification, length of stay and mortality were mentioned and verified by the operating surgical team.

Data was maintained electronically by the surgical team. Data was also entered in MS-EXCEL at the time of patient discharge. Since data was maintained on everyday basis till patient discharge and does not include follow-ups, there are no missing data.

Upon completion of study, all data will be exported to SPSS and analyzed accordingly using means, SDs, Chi-square and Fisher exact test.

ELIGIBILITY:
Inclusion Criteria:

* 1. All patients who underwent major gastrointestinal surgery and received perioperative TPN or postoperative TPN

Exclusion Criteria:

* Perioperative TPN administration that did not follow the study protocol
* TPN given for reasons other than malnutrition

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients presenting to the Surgery department at Nepal Medical College teaching hospital and having malnutrition.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
studying the effects of TPN on length of hospital stay | through study completion, an average of 5years
  comparison of perioperative and postoperative TPN in terms of mean length of stay in days
studying the effects of TPN on mortality | through study completion, an average of 5years
  comparison of perioperative and postoperative TPN in terms of number of mortality cases
studying the effects of TPN on complications using grades | through study completion, an average of 5years
  comparison of perioperative and postoperative TPN in terms of Clavien-Dindo classification grades
studying the effect of albumin levels on length of hospital stay | through study completion, an average of 5years
  comparison of low and normal albumin levels in terms of mean length of stay in days
studying the effect of albumin levels on mortality | through study completion, an average of 5years
  comparison of low and normal albumin levels in terms of number of mortality cases
studying the effect of albumin levels on complication using grades | through study completion, an average of 5years
  comparison of low and normal albumin levels in terms of Clavien-Dindo Classification grades

CONTACTS AND LOCATIONS:
Locations (1):
- Nepal Medical College Teaching Hospital, Kathmandu, Bagmati, Nepal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jensen GL, Mirtallo J, Compher C, Dhaliwal R, Forbes A, Grijalba RF, Hardy G, Kondrup J, Labadarios D, Nyulasi I, Castillo Pineda JC, Waitzberg D; International Consensus Guideline Committee. Adult starvation and disease-related malnutrition: a proposal for etiology-based diagnosis in the clinical practice setting from the International Consensus Guideline Committee. JPEN J Parenter Enteral Nutr. 2010 Mar-Apr;34(2):156-9. doi: 10.1177/0148607110361910. PMID 20375423
- [Background] Thomas MN, Kufeldt J, Kisser U, Hornung HM, Hoffmann J, Andraschko M, Werner J, Rittler P. Effects of malnutrition on complication rates, length of hospital stay, and revenue in elective surgical patients in the G-DRG-system. Nutrition. 2016 Feb;32(2):249-54. doi: 10.1016/j.nut.2015.08.021. Epub 2015 Sep 25. PMID 26688128
- [Background] Lakananurak N, Gramlich L. The Role of Preoperative Parenteral Nutrition. Nutrients. 2020 May 6;12(5):1320. doi: 10.3390/nu12051320. PMID 32384662
- [Background] Zhao XF, Wu N, Zhao GQ, Liu JF, Dai YF. Enteral nutrition versus parenteral nutrition after major abdominal surgery in patients with gastrointestinal cancer: a systematic review and meta-analysis. J Investig Med. 2016 Jun;64(5):1061-74. doi: 10.1136/jim-2016-000083. Epub 2016 Apr 25. PMID 27112357

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-21): https://cdn.clinicaltrials.gov/large-docs/32/NCT06573632/Prot_SAP_000.pdf